CLINICAL TRIAL: NCT04394806
Title: The Early and Late Contribution of Fasting and Postprandial Triglycerides on Newborn Subcutaneous and Intrahepatic Fat in Pregnancy
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0706
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Pregnancy
Keywords: Triglycerides; Glucose; Adiposity; Air displacement plethysmography; Continuous glucose monitoring
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, cord blood, cord and placental tissue,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study plans to learn more about how triglyceride levels in pregnancy affect newborn fat mass. Obesity in pregnancy, in the absence of gestational diabetes, is now the most common cause of large-for-gestational-age infants and increased newborn fat mass. Previous data supports the idea that maternal triglycerides, not glucose, are the strongest predictor of both total newborn fat mass and liver fat. In this study, mothers will monitor triglyceride and glucose levels at specific points in pregnancy using point-of-care meters at home. Two weeks after birth, infants will have total fat measured by air-displacement plethysmography (PEAPOD) and liver fat measures by Magnetic Resonance Spectroscopy (MRS). The central hypothesis is that in obesity, fasting triglycerides and postprandial triglycerides will predict newborn fat mass in a free-living environment.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women less than 16 weeks gestational age
* Between the ages of 21-39 years
* Pre-pregnancy BMI 28-39 kg/m2

Exclusion Criteria

* Pre-gestational diabetes or prediabetes
* History of gestational diabetes
* History of pre-eclampsia, spontaneous pre-term delivery, or gestational hypertension <34wks
* Tobacco or illicit substance use
* Chronic steroid use

Ages: 0 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Overweight and obese pregnant women between the ages of 20-39 years old, who are receiving care at a University of Colorado Health Facility.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Newborn Fat Mass | 7-14 days after birth
  Newborn fat mass measured by air displacement plethysmography (PeaPod)

SECONDARY OUTCOMES:
Newborn Intrahepatic Fat | 7-14 days after birth
  Newborn intrahepatic fat measured by Magnetic Resonance Spectroscopy (MRS)

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Barbour, MD, MSPH, Principal Investigator — University of Colorado, Denver; Teri L Hernandez, PhD, RN, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado/Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbour LA, Farabi SS, Friedman JE, Hirsch NM, Reece MS, Van Pelt RE, Hernandez TL. Postprandial Triglycerides Predict Newborn Fat More Strongly than Glucose in Women with Obesity in Early Pregnancy. Obesity (Silver Spring). 2018 Aug;26(8):1347-1356. doi: 10.1002/oby.22246. Epub 2018 Jun 22. PMID 29931812